CLINICAL TRIAL: NCT00976976
Title: Phase 2 Study of Adjuvant Chemotherapy With Docetaxel, Capecitabine and Cisplatin in Patients With Advanced Gastric Cancer
Brief Title: Adjuvant Chemotherapy With Docetaxel, Capecitabine and Cisplatin in Patients With Advanced Gastric Cancer: Adjuvant DXP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC0604
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Resected Advanced Gastric Cancer
Keywords: Resected advanced gastric cancer stage IIIB and IV
MeSH Terms: interventions — Docetaxel; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DXP (Experimental)
  Interventions: Drug: docetaxel, capecitabine, cisplatin

INTERVENTIONS:
Drug: docetaxel, capecitabine, cisplatin — Docetaxel 60 mg/m2 IV (day 1) every 21 days capecitabine 1,875 mg/m2/day PO, divided two (day 1-day14) every 21 days Cisplatin 60 mg/m2 IV (day 1) every 21 days
  Other Names: docetaxel,xeloda,cisplatin

SUMMARY:
Despite the improvement of surgical resection as primary curative treatment for gastric cancer, more than 70% of patients with stage IIIB and IV disease undergoing radical primary tumor resection relapse and die within 5 years. Therefore, there is an urgent need to further improve the treatment for gastric cancer in this population. Recently reported phase III study comparing capecitabine/cisplatin (XP) versus 5-FU/cisplatin (FP), XP showed better activity and tolerability compared with FP. To improve treatment outcomes of XP chemotherapy, the investigators performed a phase I-II study of docetaxel, capecitabine and cisplatin in advanced gastric cancer (AGC). Phase I-II study of docetaxel, capecitabine and cisplatin as first-line chemotherapy in advanced gastric cancer (Kang et al, Proc Am Soc Clin Oncol 22,328.2003). The docetaxel/capecitabine/cisplatin (DXP) chemotherapy was highly active for the 1st-line chemotherapy of AGC. These findings and experience encourages the investigators to design the adjuvant trial of DXP chemotherapy in patients with resected gastric cancer. The aim of this study is to assess the efficacy and safety of adjuvant DXP in this patient population.

DETAILED DESCRIPTION:
Previous in phase II study of docetaxel, capecitabine and cisplatin,total 40 pts with measurable disease, median 6 cycles of chemotherapy, there were 4 confirmed complete responses (CRs) and 23 confirmed partial responses (PRs), with the overall response rate of 67.5% (95% confidence interval, 52.7 ~ 82.3) in intention-to-treat analysis. Ten patients underwent surgical resection after 4 ~ 9 cycles of chemotherapy. Four pathologic CRs were identified. With a median follow-up of 14 months (range, 1 to 28), median time to progression was 7.7 months, and median overall survival was 16.9 months. The DXP chemotherapy was highly active for the 1st-line chemotherapy of AGC (Kang et al, Proc Am Soc Clin Oncol 22,328.2003).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented gastric adenocarcinoma
* Age 18 -70
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Pathologic stage IIIB or IV
* complete resection (R0 resection)

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* R1 or R2 resection
* Presence of distant metastasis
* Gastric outlet obstruction or intestinal obstruction
* Evidence of gastrointestinal bleeding
* Other serious illness or medical conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
This protocol will evaluate the possible benefit of adjuvant docetaxel, capecitabine, and cisplatin combination chemotherapy in patients with resected gastric cancer pathologic stage IIIB and IV in terms of relapse free survival. | 5 years

SECONDARY OUTCOMES:
Investigate the safety profiles, patient tolerance, and overall survival in this population | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea